CLINICAL TRIAL: NCT03662841
Title: Ablative Chemoembolization for Unresectable and Large Hepatocellular Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor patient accrual
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon Yu, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIR-18-08
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2022-02

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Use of ACE for HCC of size > 10cm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACE for HCC of size >10cm (Other): Ablative chemoembolization (ACE) using Lipiodol-ethanol and anhydrous cisplatin
  Interventions: Procedure: Ablative chemoembolization (ACE)

INTERVENTIONS:
Procedure: Ablative chemoembolization (ACE) — Ablative chemoembolization (ACE) using Lipiodol-ethanol and anhydrous cisplatin

SUMMARY:
The objective of this study is to study the safety and tumor response of ACE for large HCC.

DETAILED DESCRIPTION:
Transarterial treatment has been playing an important role in the treatment algorithm for patients with multifocal or large intrahepatic hepatocellular carcinoma not eligible for surgical resection, transplantation, or local ablative therapy. Among the patient group with intermediate tumor stage, in which the tumor dimension exceeds 10cm, the treatment outcome of conventional chemoembolization (cTACE), chemoembolization using drug eluting beads (DEB-TACE) and radioembolization using yttrium 90 is generally unsatisfactory. Some would consider HCC of size >10cm a relative contraindication for cTACE because of the poor treatment outcome. However, there is no better alternative treatment for local control of these tumors. Ablative chemoembolization (ACE) using Lipiodol-ethanol and anhydrous cisplatin has been found to be highly effective for local control of HCC as compared to cTACE in a case-control study. It is hypothesized that ACE is safe and effective for local control of large HCC of size >10cm.

ELIGIBILITY:
Inclusion Criteria:

1. Signage of a written informed consent
2. Age above 18 years
3. HCC unsuitable for resection
4. Child-Pugh A or B cirrhosis
5. Eastern Cooperative Oncology Group performance score 0 or 1
6. No previous treatment with liver resection, ablation, chemotherapy, radiotherapy or transarterial embolization (with or without chemotherapy),
7. HCC diagnosed by typical enhancement patterns on cross sectional imaging or histology.
8. No extra-hepatic involvement on non-enhanced CT thorax and triphasic contrast enhanced CT abdomen.
9. No invasion of portal vein or hepatic vein
10. Massive expansive tumor morphology with measurable lesion on CT (characterized by well-defined spherical or globular configuration, with or without tumor capsule or satellite lesions)
11. Total tumor mass < 50% liver volume
12. Size of any individual tumor >10cm in largest dimension

Exclusion Criteria:

1. History of acute tumor rupture presenting with hemo-peritoneum
2. Biliary obstruction not amenable to percutaneous or endoscopic drainage
3. Child-Pugh C cirrhosis
4. History of hepatic encephalopathy
5. Intractable ascites not controllable by medical therapy
6. History of variceal bleeding within last 3 months
7. Serum total bilirubin level > 50 umol/L
8. Serum albumin level < 25g/L
9. INR > 1.7
10. Serum creatinine level > 150 mmol/L.
11. Infiltrative tumor morphology (characterized by ill- defined tumor margin and amorphous configuration) or diffuse tumor morphology (characterized by large number of small nodules)
12. Arterio-portal venous shunt affecting >1 hepatic segment on CT
13. Arterial-hepatic venous shunt with hepatic vein opacified in arterial phase on CT

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Time to progression | 3 to 6 months after treatment
  the interval between the first treatment date and the date of radiological progression, including intralesional progression, extralesional progression, or extra-hepatic progression

SECONDARY OUTCOMES:
Tumor response | 3 to 6 months after treatment
  Tumor response at 3 month and 6 month from the date of first treatment as evaluated by triphasic contrast enhanced CT according to the EASL criteria

CONTACTS AND LOCATIONS:
Overall Officials: Simon Yu, Principal Investigator — DIIR, CUHK, Hong Kong
Locations (1):
- Department of Imaging and Interventional Radiology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong